CLINICAL TRIAL: NCT06767566
Title: Ketamine Pharmacokinetics and Pharmacodynamics for Postpartum Depression and Pain After Cesarean Delivery
Acronym: PREPARE-2
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Grace Lim, MD, MS (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Grace Lim, MD, MS, Associate Professor, Chief Obstetric & Women's Anesthesiology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY22100019; R01MH134538 (NIH)
Record Dates: First submitted 2024-11-21; First posted 2025-01-10 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Pain; Postpartum Depression
Keywords: Cesarean Delivery
MeSH Terms: conditions — Pain; Depression, Postpartum | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: 20 subjects will be cesarean delivery population 30 subjects will be Healthy Control population (N=15 nonpregnant female, N=15 male) Both groups will receive same intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ketamine Infusion: Cesarean Delivery Population (Experimental): Loading dose infusion for 1 hour followed immediately by maintenance dose infusion for 11 hours.
  Interventions: Drug: Ketamine (Ketalar)
- Ketamine Infusion: Healthy Control Population (Experimental): Loading dose infusion for 1 hour followed immediately by maintenance dose infusion for 11 hours.
  Interventions: Drug: Ketamine (Ketalar)

INTERVENTIONS:
Drug: Ketamine (Ketalar) — Loading Dose: 0.18 mg/kg/hr x 1 hour; Maintenance Dose 0.05 mg/kg/hr x 11 hours
  Other Names: 0.18 mg/kg/1hr loading dose Ketamine

SUMMARY:
The purpose of this study is to identify pharmacokinetics of postpartum ketamine infusion. This study will assess ketamine kinetics and metabolism in this setting. Ketamine is expected to exert different kinetics during the physiologic state of post-pregnancy. The goal in conducting this study is to better understand the pharmacokinetics and pharmacodynamics of postpartum ketamine infusion. A secondary goal is to compare these kinetics to reproductive age matched controls and to assess sex differences in ketamine pharmacokinetics.

The peripartum group of this study will receive ketamine after cesarean delivery, while the control group will consist of non-pregnant female subjects and male subjects receiving the same infusion protocol.

DETAILED DESCRIPTION:
A lack of data on new pain treatments in pregnancy puts 1.2 million US women having cesarean delivery (CD) every year at risk for poor pain control, depressed mood, and poor recovery. Evidence of successful post-surgical pain management and rapid reduction of depressive symptoms render ketamine a great candidate for post-CD pain management and potential reduction of postpartum depression (PPD) symptomology. Knowledge gaps in ketamine pharmacokinetics (PK) in the postpartum period limit an informed approach to its use for postpartum analgesia and PPD mitigation strategies. Similarly, knowledge gaps about sex differences in ketamine PK limit understandings about potential heterogeneity of treatment effects. This study aims to better understand the pharmacokinetics and pharmacodynamics of ketamine in postpartum women. Secondarily, it will assess key differences in postpartum ketamine PK compared to non-pregnant female controls. Secondarily it will assess key sex differences in ketamine metabolism between male and female subjects.

Peripartum females undergoing cesarean delivery will receive a ketamine infusion for 12 hours after cord clamping. Samples will be taken to characterize ketamine PK (primary objective). Healthy volunteer control females and males will receive the same ketamine infusion dosing schematic. Comparisons will be made between peripartum females and non-pregnant female controls, and between female and male controls (secondary objectives).

ELIGIBILITY:
Peripartum Participants:

Inclusion Criteria

* Cesarean delivery
* Adults 18 years and older
* Term delivery ≥ 37 weeks gestation anticipated at time of delivery
* ASA PS 2 or 3
* Able to provide informed consent
* One of the following must be met for inclusion: Not planning to breastfeed OR ketamine use indicated for pain management plan.

Exclusion Criteria

* Patient going under general anesthesia for cesarean delivery
* Allergy to study medication (ketamine)
* ASA PS 4 +
* Contraindications to neuraxial anesthesia
* Preterm delivery (<37 weeks gestation)
* Anticipated fetal-neonatal complex care plan as indicated in the patient's chart
* Patient history of ketamine or PCP abuse
* Patient history of schizophrenia or psychosis
* Patient history of liver or renal insufficiency
* Patient history of uncontrolled hypertension, chest pain, arrhythmia, head trauma, or intracranial hypertension, uncontrolled hyperthyroidism, or other contraindications to ketamine
* Participating in another pain or depression intervention trial
* Undergoing hormonal or gender affirming therapies
* Pre-eclampsia with severe features
* Hemodynamic instability
* Inability to participate in study procedures for any reason
* Contraindicated medications use: oral antihypertensive medications (exclusion: hypertensive disorders of pregnancy), intravenous magnesium (exclusion: pre-eclampsia with severe features), ketamine/phencyclidine/psilocybins/any other psychedelics (exclusion: ketamine or PCP abuse), lithium/valproate/carbamazepine/lamotrigine/haloperidol/chlorpromazine/fluphenazine/aripiprazole/clozapine/other typical or atypical antipsychotic medications (exclusion: schizophrenia or psychosis)

Control Participants

Inclusion Criteria

* Age 18 years and older
* Sex: Male or Female
* Able to provide informed consent
* ASA PS 1, 2, or 3

Exclusion Criteria

* Allergy to study medication (ketamine)
* ASA PS 4 +
* Inability to participate in study procedures for any reason
* Patient history of ketamine or PCP abuse
* Patient history of schizophrenia or psychosis
* Patient history of liver or renal insufficiency
* Patient history of uncontrolled hypertension, chest pain, arrhythmia, head trauma, intracranial hypertension, uncontrolled hyperthyroidism, or other contraindications to ketamine
* Participating in another pain or depression intervention trial
* Hemodynamic instability
* Pregnant or pregnant within the last 6 weeks
* Unwilling to provide urine sample for pregnancy testing (female controls)
* Undergoing hormonal or gender affirming therapies
* Contraindicated medications use: ketamine, phencyclidine, psilocybins, or other psychedelics (exclusion: ketamine or PCP abuse), lithium/valproate/carbamazepine/lamotrigine/haloperidol/chlorpromazine/fluphenazine/aripiprazole/clozapine, or other typical or atypical antipsychotic medications (exclusion: schizophrenia or psychosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2027-12-07 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Maternal ketamine area under the curve (AUC) | 0 to 24 hours from initiation of ketamine infusion
  Ketamine area under the plasma concentration-time curve (AUC 0-∞) (AUC, mcg*min/mL), which reflects the actual body exposure to ketamine after administration of ketamine.

SECONDARY OUTCOMES:
Patient reported acceptability of any reported side effects | 0 to 24 hours after initiation of ketamine infusion
  Proportion (%) of patient cohort reporting acceptability of ketamine infusion
Pain area under the curve (AUC) | 0 to 24 hours after initiation of ketamine infusion
  Pain score area under the curve (AUC) where pain scores are measured from 0 (no pain) to 10 (worst imaginable pain), for the duration of epidural analgesia.
Depression scores (Peripartum) | Baseline to week 12 post-infusion
  Depression scores as defined by the Edinburgh Postnatal Depression Scale (Peripartum Group), scale 0-30, measured among the peripartum cohort.
Depression Scores (control) | Baseline to week 12 post-infusion
  Depression scores as defined by the Patient Health Questionnaire (PHQ-9) (Control Group), scale 0-27, measured among the control nonperipartum cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Grace Lim, MD, MSc, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Magee Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - UPMC Montefiore Clinical and Translational Research Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be available for public benefit and knowledge. Items for uploading will include clinical measures, patient reported outcomes, psychometric testing data, sensory testing data, and all PK data. Technical protocols and any other data collected under this project will be shared upon request to allow others to perform secondary analyses.
Supporting Information: Study Protocol, CSR
Time Frame: Beginning with 3 months and ending at 5 years following article publication.
Access Criteria: Researchers who propose a methodologically sound proposal may submit said proposals to limkg2@upmc.edu. To gain access to data, requestors will need to sign a data access agreement.